CLINICAL TRIAL: NCT04230668
Title: A Pilot Effectiveness Trial of Cognitive Processing Therapy Augmented With Suicide Risk Management for Individuals With Comorbid PTSD and BPD
Brief Title: Cognitive Processing Therapy (CPT) for Posttraumatic Stress Disorder and Borderline Personality Disorder (PTSD-BPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Palo Alto University (Other)
Collaborators: Toronto Metropolitan University (Other); York University (Other); Stanford University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Janice Kuo, Professor, Palo Alto University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPT for PTSD-BPD; 1R34MH124968-01A1 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Posttraumatic Stress Disorder; Borderline Personality Disorder
Keywords: Cognitive Processing Therapy; Suicide Risk Management; Suicide; Self-harm
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Borderline Personality Disorder; Suicide; Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a two-phased study. Phase 1 of this investigation will consist of an initial case series in which the CPT+SRM manual will be developed along with fidelity measures. The finalized treatment manual will then be tested in Phase 2, a randomized-controlled trial comparing 12 individual sessions/6 weeks of CPT+SRM versus 6 weeks of TAU+SRM.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPT + SRM (Experimental): Participants will be randomized to teletherapy sessions of Cognitive Processing Therapy + Suicide Risk Management for PTSD-BPD which will be administered twice weekly over 6 weeks, for a total of 12 sessions.
  Interventions: Behavioral: Cognitive Processing Therapy with Suicide Risk Management
- TAU + SRM (Experimental): Participants will be randomized to teletherapy sessions with only Suicide Risk Management for PTSD-BPD which will be administered once a week for 6 weeks, for a total of 6 sessions.
  Interventions: Behavioral: Treatment as Usual with Suicide Rick Management

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy with Suicide Risk Management — CPT is an evidence-based treatment for PTSD. This first-line treatment for PTSD will be adapted and combined with SRM into 12 sessions, 60-90 minutes targeting both PTSD and BPD. Individuals assigned to this intervention will attend treatment sessions, and be asked to do treatment homework at home. The primary outcomes are PTSD and BPD severity.
  Arms: CPT + SRM
Behavioral: Treatment as Usual with Suicide Rick Management — In the Suicide Risk Management only condition, participants will receive 6 weekly sessions over the course of six weeks focused on suicide stabilization and management. Each SRM session will be variable lengths, depending on the participants' suicide risk and can be up to 60 minutes.
  Arms: TAU + SRM

SUMMARY:
Posttraumatic Stress Disorder (PTSD) with co-occurring Borderline Personality Disorder (BPD) (i.e., PTSD-BPD) is common (as high as 58%), debilitating, costly, and limited treatment options available for this population. PTSD-BPD is associated with even greater functional impairment and higher healthcare burden than either disorder alone. There are surprisingly few treatments available for this clinical profile, despite its association with major negative health outcomes, cost, and morbidity. There is a pressing need to innovate treatments that can effectively and efficiently treat PTSD-BPD. The existing treatments used for PTSD-BPD are lengthy, laborious, resource-intensive, and require complete cessation of suicidal behaviors prior to treatment. Furthermore, no integrated treatment has been innovated to deliver the active ingredients to efficiently affect the mechanisms underpinning this comorbidity. The investigators propose to examine an adapted version of a first-line PTSD intervention, Cognitive Processing Therapy, augmented with a Suicide Risk Management, i.e., (CPT+SRM) as a brief (12 sessions) and more parsimonious treatment alternative that strategically targets shared mechanisms underpinning PTSD and BPD. The purpose of this pilot study is to 1) collect initial feasibility, acceptability, and safety data on this adapted treatment, 2) conduct a pilot randomized clinical trial evaluating the efficacy of CPT+SRM versus Treatment as Usual (TAU) + SRM, and 3) evaluate two targets (i.e, improvements in emotional intensity and cognitive dysfunction) as mechanisms leading to change in our primary outcomes. Both treatment conditions will be administered via telehealth.

Potential benefits include reduction in participants' PTSD, BPD and other mental health symptoms. Additionally, this work could benefit the community by improving the treatment repertoire for PTSD-BPD. Potential risks include emotional distress, suicidality, and/or self-harm. Participants may experience discomfort and/or distress while discussing participants trauma(s) and mental health. These risks will be mitigated using a suicide risk management protocol which therapists in the assessment of risk and protective factors of suicide, followed by documentation for the decision-making around the management of risk.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Must reside in the Bay Area, CA
* Current DSM-5 diagnosis of PTSD and BPD
* Must be willing to be audio- or videorecorded for assessment and treatment sessions

Exclusion Criteria:

* Acute mania, acute psychosis, or intellectual disability
* Conditions requiring medical attention to a potentially life-threatening illness (e.g., severe anorexia nervosa)
* Severe impairments in written and aural comprehension
* EU individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 30-item clinician administered structured interview based on the DSM-5 PTSD criteria.
Borderline Symptom List 23 (BSL-23) [SELF-REPORT] | Baseline, once a week while in treatment (for 6 weeks)
  A self-report measure of borderline personality disorder (BPD) severity. The measure captures subjective ratings of the following symptoms: self-perception, affect regulation, self destruction, dysphoria, loneliness, intrusions, and hostility (Bohus et al., 2009).

SECONDARY OUTCOMES:
Suicide Attempt Self-Injury Interview (SASII) | 3-weeks, Post-treatment/6-weeks, 3-month follow-up
  Assess characteristics of self-harm (i.e., suicide attempts and NSSI), including frequency, medical severity, intent to die, lethality, and precipitants of self-harm since the previous assessment.
Difficulties in Emotion Regulation Scale (DERS) [SELF-REPORT] | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A self-report measure assessing various dimensions of emotion dysregulation (Gratz & Roemer, 2004).
Posttraumatic Cognitions Inventory (PTCI) [SELF-REPORT] | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 33-item scale assessing post-traumatic symptoms, reactions and appraisals. The measure possesses three subscales; negative cognitions related to the self, negative cognitions related to the world, and self-blame cognitions related to the traumatic event.
Beck's Depression Inventory-II (BDI-II) [SELF-REPORT] | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 21-item, self-report inventory that measures the severity of depression symptomatology. It corresponds closely to DSM-5 depression criteria and is found to be a more reliable measure of depression (Beck & Steer, 1988).
State-Trait Anxiety Inventory, Trait Version (STAI-T) | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A measure that consists of 20 items for assessing trait anxiety and 20 for assessing state anxiety. It is used to diagnose anxiety and to help distinguish it from depressive syndromes.
State-Trait Anger Expression Inventory-II (STAXI-II) [SELF-REPORT] | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 57-item self-report measure that examines the expression, control, and experience of anger (Schamborg, Tully, & Browne, 2016).
Social Adjustment Scale - Self Report (SAS-SR) [SELF-REPORT] | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A measure that consists of 54 items for assessing role performance in six areas of functioning, including work, social and leisure activities, relationships with extended family, role as a marital partner (if applicable), parental role (if applicable), and role within the family unit.
Trauma-Related Guilt Inventory (TRGI) [SELF-REPORT] | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 32-item self-report measure that is designed to measure guilt experienced as a result of a traumatic event. It is composed of three subscales including; guilt cognitions, distress and global guilt.
Suicidal Behaviors Questionnaire-Revised | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  Scores range from 3 to 18, with 18 being higher suicide risk.
Substance Use Inventory (SUI) | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A brief measure with detailed questions regarding participants' use and primary route of different substances they used in the last seven days. The individuals' are also asked about the average dollar amount spent on each drug and in a single day. (Weiss, et al., 1995).
PTSD Checklist-5 (PCL-5) [SELF-REPORT] | Baseline, once a week while in treatment (for 6 weeks)
  A 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. It is used to help screen individuals for PTSD as well as monitor their symptom changes during and after treatment.
Acceptability of Intervention Measure (AIM) | Baseline and Post-treatment/6-weeks
  A 4-item measure which asks therapists and patients about their perceived acceptability of the intervention on a 5-point Likert scale.
Treatment sessions attended | Pre-post treatment (6 weeks)
  Feasibility as measured by number of treatment sessions
Rate of dropout | Pre-post treatment (6 weeks)
  Feasibility as measured by rate of treatment dropout
Emotional Reactivity and Attentional Biases via Oddball task | Baseline, Post-treatment/6-weeks, 3-months follow-up
  Used as a behavioral measure of changes in emotional reactivity and attentional biases- our two propose mechanisms of change in CPT+SRM. The oddball task is computer-based task (Hayes, et al., 2009) designed to measure emotional reactivity and attentional biases. Participants will view a pseudorandom distribution of brief presentations of emotionally-salient distractors (negative images depicting mutilations, burn victims, attacks, sick individuals), neutral distractors (matched with negative images for luminance, presence of human figures, chromatic features), baseline standards (squares), and attention "targets" (circles) in an event-related design. Participants will be instructed to press the same button for all stimuli, but a different button for attention targets. Behavioral changes associated with emotional reactivity and attention bias will be assessed using response latency and accuracy scores for emotional and attention targets, respectively.
Mental Health Involvement Scale [SELF-REPORT] | Post-treatment/6-weeks
  A 9-item measure used to inquire about other ancillary services (e.g., group treatment, couples/family therapy) that participants are receiving throughout the study. This is a measure developed and used in prior research by the investigative team, but currently does not have published psychometric properties.
Measure of CPT+SRM Uptake [SELF-REPORT] | 9-months after concluding treatment with the last study participant
  Measures uptake of the treatment using an adapted measure from LoSavio, et al. (2019). This brief survey will assess clinicians' ongoing use of CPT+SRM since their participation in the study (e.g., whether they continue to offer CPT+SRM, the number of clients they have offered CPT+SRM to, average number of sessions attended, etc.) and further inform whether our training methods and treatment will have a lasting impact on practice approaches in community settings. There are no psychometric data available for this questionnaire.
Unanticipated Problems Involving Risk to Subjects or Others (UPIRSO) | Baseline, 3-weeks, Post-treatment/6-weeks
  Safety of the treatment will be monitored via unanticipated problems involving risk to subjects or others (UPIRSO) that occur throughout treatment and the number of mental health hospitalizations.
The International Personality Disorder Exam (IPDE, BPD only) | Baseline
  A well-established diagnostic instrument used by the World Health Organization, will be used to identify the presence and severity of BPD. The IPDE also allows for a dimensional assessment of BPD.
The Structured Clinical Interview for the Diagnostic and Statistical Manual-5 (SCID-5) | Baseline
  Used to obtain other DSM-5 diagnoses.
The Lifetime Suicide Attempt Self-Injury Interview (L-SASII) | Baseline
  A semi-structured interview, will assess characteristics of self-harm (i.e., suicide attempts and NSSI), including frequency, medical severity, intent to die, lethality, and precipitants of self-harm.
A Demographic Form [SELF-REPORT] | Baseline
  Used in previous PTSD treatment studies will also be used to measure a range of demographic data.
Trauma-Related Shame Inventory (TRSI) [SELF-REPORT] Trauma-Related Shame Inventory (TRSI) [SELF-REPORT]: is a 24-item self-report measure that evaluates levels of shame in the context of one's trauma. -- | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 24-item self-report measure that evaluates levels of shame in the context of one's trauma.
Patient Health Questionnaire - 9 (PHQ-9) | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 9-item self-report measure that evaluates severity of depression symptoms.
Generalized Anxiety Disorder - 7 (GAD7) | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 7-item self-report measure that evaluates severity of generalized anxiety symptoms.
WHO Disability Assessment Schedule (WHODAS) 2.0 (12-Item Version) | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 12-item self-report measure of disability across six domains (understanding and communicating, getting around, self-care, getting along with people, life activities, and participation in society).
DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure-Adult | Baseline, 3-weeks, Post-treatment/6-weeks, 3-months follow-up
  A 23-item self-report measure of psychiatric symptoms that cut across diagnostic categories.

CONTACTS AND LOCATIONS:
Overall Officials: Janice R Kuo, PhD, Principal Investigator — Palo Alto University
Locations (1):
- Palo Alto University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resick, P. A., Monson, C. M., & Chard, K. M. (2016). Cognitive processing therapy for PTSD: A comprehensive manual. New York, NY: Guilford Press.
- [Background] Stanley, B., & Brown, G. (2012). Safety planning intervention: A brief intervention to mitigate suicide risk. Cognitive and Behavioural Practice, 19(2), 256-264.